CLINICAL TRIAL: NCT04686175
Title: A Phase 1/2, Open-Label, Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of INZ-701 Followed by an Open-Label Long-Term Extension Period in Adults With ENPP1 Deficiency
Brief Title: Evaluation of Safety, Tolerability, and Efficacy of INZ-701 in Adults With ENPP1 Deficiency
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Inozyme Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INZ701-101; 2020-003716-27 (EudraCT Number)
Record Dates: First submitted 2020-12-22; First posted 2020-12-28 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Ectonucleotide Pyrophosphatase/phosphodiesterase1 Deficiency; Autosomal Recessive Hypophosphatemic Rickets; Generalized Arterial Calcification of Infancy
Keywords: ectonucleotide pyrophosphatase/phosphodiesterase1 deficiency; hypopyrophosphatemia; ENPP1; Generalized Arterial Calcification of Infancy; GACI; Autosomal Recessive Hypophosphatemic Rickets Type 2; ARHR2
MeSH Terms: conditions — Hypophosphatemic Rickets, Autosomal Recessive, 1; Arterial calcification of infancy

STUDY DESIGN:
Intervention Model Description: Study INZ701-101 is a Phase 1/2, multi-center, open-label, first-in-human (FIH), multiple ascending dose (MAD) study followed by a long-term open-label extension period conducted in adults with ENPP1 Deficiency. The study design during the Dose Evaluation Period is a MAD 3+3 with 3 dose cohorts.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- INZ-701 (Experimental): The study design of the Dose Evaluation Period is a MAD 3 + 3 with 3 dose cohorts. Additional cohorts may be added to evaluate an intermediate dose and/or an alternative dosing regimen of an existing dose level.
  Based on nonclinical findings and nonclinical pharmacology modeling, the initial planned doses will be 0.2 mg/kg, 0.6 mg/kg, and 1.8 mg/kg all twice weekly, not to exceed 3.6 mg/kg weekly.
  During the Extension Period, visits will be every 4 weeks until Week 48 and then every 12 weeks until the subject leaves the study. Subjects will complete an End of Study (EOS) Visit (Safety Follow-up Visit) 30 days after their last dose of INZ-701 (greater than 5 half-lives of INZ-701) for all subjects.
  Interventions: Drug: INZ-701

INTERVENTIONS:
Drug: INZ-701 — INZ701-101 is a recombinant fusion protein that contains the extracellular domains of human ENPP1 coupled with an Fc fragment from an immunoglobulin gamma-1 (IgG1) antibody.
  Other Names: rhENPP1-Fc

SUMMARY:
The purpose of this study is to assess the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of multiple ascending doses of INZ-701, an ectonucleotide pyrophosphatase/phosphodiesterase 1 (ENPP1) enzyme replacement therapy, for the treatment of ENPP1 Deficiency. The goal of the study is to identify a dose regimen for further clinical development in the treatment of ENPP1 Deficiency.

DETAILED DESCRIPTION:
INZ-701 is an ectonucleotide pyrophosphatase/phosphodiesterase 1 (ENPP1) enzyme replacement therapy (ERT) in development for the treatment of ENPP1 Deficiency, an ultra-rare genetic disorder with an incidence of 1 in 64,000 pregnancies.

Study INZ701-101 is a Phase 1/2, multicenter, open-label, FIH, MAD, dose-finding study followed by a long-term open-label Extension Period conducted in adults with ENPP1 Deficiency. This study is designed to assess the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of multiple ascending doses of INZ-701. The goal of the study is to identify a dose and dose schedule (number of doses per week) for further clinical development. No placebo will be used in the study. Subjects will be 18 to <65 years of age, with a confirmed genetic diagnosis of ENPP1 Deficiency and biochemical evidence of hypopyrophosphatemia (ie, PPi <1300 nM). Exploratory endpoints for the Extension Period of the study include evaluations of skeletal assessment (X-ray and DEXA), arterial and organ calcification (either Na18F-PET/CT or low dose CT [full body] without contrast, echocardiogram, and renal ultrasound), and cardiovascular function (echocardiogram) as well as patient reported outcomes.

Subject participation consists of a Screening Period of up to 30 days, a 32-day Dose Evaluation Period, and an Extension Period during which subjects may continue to receive INZ-701 (with options for self-, caregiver-, or healthcare provider administration) until INZ-701 is approved and available in the country where the subject resides or until an alternative study for subjects to continue receiving study drug is available. During the Extension Period, follow-up visits will be conducted every 4 weeks until Week 48, followed by every 12 weeks until the subject leaves the study.

Subjects will complete an End of Study (EOS) Visit (Safety Follow-Up Visit) 30 days after their last dose of INZ-701.

ELIGIBILITY:
Individuals eligible to participate must meet all of the following inclusion criteria:

1. Must provide written or electronic consent after the nature of the study has been explained, and prior to any research-related procedures, per International Conference on Harmonisation (ICH) Good Clinical Practice (GCP)
2. Clinical diagnosis of ENPP1 Deficiency supported by prior identification of biallelic ENPP1 mutations (ie, homozygous or compound heterozygous)
3. Male or female, 18 to <65 years of age at Screening
4. PPi <1300 nM at Screening
5. Women of child-bearing potential (WOCBP as defined in Clinical Trials Facilitation and Coordination Group [CTFG 2020]) must have a negative serum pregnancy test at Screening
6. WOCBP and partners of fertile males who are WOCBP must be using or agree to use 1 highly effective form of contraception (per CTFG 2020) and a barrier method from at least 1 month before the first dose of INZ-701 through 30 days after the last dose of INZ-701 (greater than 5 half-lives of INZ-701). WOCBP and partners of fertile males who are WOCBP must also agree to not donate ova from the period following the first dose of INZ-701 through 30 days after last dose of INZ-701.
7. Males who are sexually active must agree to use condoms from the period following first dose of INZ-701 through 30 days after the last dose of INZ-701. Males must also agree to not donate sperm from the period following the first dose of INZ-701 through 30 days after last dose of INZ-701.
8. In the opinion of the Investigator, must be willing and able to complete the Dose Evaluation Period.
9. Agree to provide access to relevant medical records.

Individuals who meet any of the following exclusion criteria will not be eligible to participate:

1. In the opinion of the Investigator, presence of any clinically significant disease (outside of those considered associated with the diagnosis of ENPP1 Deficiency) that precludes study participation or may confound interpretation of study results, including known uncontrolled cardiovascular, thyroid disease, or unrelated connective tissue, bone, mineral, lipid, or muscle disease
2. Clinically significant abnormal laboratory result at Screening in the opinion of the Investigator, including but not limited to screening laboratory results demonstrating

   1. estimated glomerular filtration rate (eGFR) (Chronic Kidney Disease-Epidemiology Collaboration [CKD-EPI] equation) < 60 mL/min/1.73m^2,
   2. 25-hydroxyvitamin D (25[OH]D) levels <12 ng/mL, or
   3. Intact parathyroid hormone (PTH) >40% above the upper limit of normal
3. Known active fungal, bacterial, and/or viral infection including human immunodeficiency virus, hepatitis B virus, hepatitis C virus, or COVID-19 virus. In Germany and France, a negative COVID-19 test result is required within 5 days prior to the first dose of INZ-701.
4. Malignancy within the last 5 years, except non-melanoma skin cancers or cervical carcinoma in situ
5. Known intolerance to INZ-701 or any of its excipients
6. Unable or unwilling to discontinue the use of any prohibited medication (examples include 1,25-dihydroxy vitamin D, phosphate, anti-FGF23 [eg, burosumab], calcimimetics, calcium-containing antacids, systemic corticosteroids, PTH suppressors). Discontinuation should be undertaken only if considered not detrimental and indicated by the subject's treating physician.
7. Concurrent participation in another non-Inozyme interventional clinical study and/or receipt of any other investigational new drug within 5 half-lives of the last dose of the other investigational product or from 4 weeks prior to the first dose of INZ-701, whichever is longer, or use of an investigational device, through completion of participation in the study
8. Subjects who are pregnant, trying to become pregnant, or breastfeeding
9. Subjects who are trying to father a child

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2021-11-21 (Actual); Primary Completion 2024-10-29 (Actual); Study Completion 2024-12-13 (Actual)

PRIMARY OUTCOMES:
Number of Treatment Emergent Adverse Events (TEAEs) | 32 days (Dose Evaluation Period)
  Treatment-emergent AEs are defined as any AE occurring from the first dose of INZ-701 through 30 days after the last dose of INZ-701.
Number of Treatment Emergent Adverse Events (TEAEs) | 52 weeks (Day 1 through Safety Follow-up Visit)
  Treatment-emergent AEs are defined as any AE occurring from the first dose of INZ-701 through 30 days after the last dose of INZ-701.
Incidence of Anti-Drug Antibodies (ADA) | 32 days (Dose Evaluation Period)
  For each subject, the presence of ADAs will be assessed and, if present, further evaluation will determine specificity and subtypes.
Incidence of Anti-Drug Antibodies (ADA) | 52 weeks (Baseline through Safety Follow-up Visit)
  For each subject, the presence of ADAs will be assessed and, if present, further evaluation will determine specificity and subtypes.
Area under the Plasma Concentration versus Time Curve (AUC) of INZ-701 | 32 days (Dose Evaluation Period)
  For each subject, variation of concentration of INZ-701 in the plasma will be measured via a series of blood samples obtained throughout the study, comparing the subject's baseline value over time.
Maximum Plasma Concentration (Cmax) of INZ-701 | 32 days (Dose Evaluation Period)
  For each subject, the maximum concentration of INZ-701 in the plasma will be measured via a series of blood samples obtained throughout the study, comparing the subject's baseline value over time.
Systemic Clearance of INZ-701 | 32 days (Dose Evaluation Period)
  For each subject, clearance of INZ-701 from the body will be measured via a series of blood samples obtained throughout the study, comparing the subject's baseline value over time.
Change from Baseline in Plasma Inorganic Pyrophosphate (PPi) Levels | 32 days (Dose Evaluation Period)
  For each subject, plasma PPi will be measured via a series of blood samples obtained throughout the study, comparing the subject's baseline value over time.
Change from Baseline in Plasma Inorganic Pyrophosphate (PPi) Levels | 52 weeks (Baseline through Safety Follow-up Visit)
  For each subject, plasma PPi will be measured via a series of blood samples obtained throughout the study, comparing the subject's baseline value over time.

CONTACTS AND LOCATIONS:
Overall Officials: Kurt Gunter, MD, Study Director — Inozyme Pharma, Inc.
Locations (7):
- United States (2):
  - Mayo Clinic, Rochester, Minnesota
  - Clinilabs Drug Development Corporation, Eatontown, New Jersey
- University of Saskatchewan, Saskatoon, Saskatchewan, Canada
- Necker University Hospital-Sick Children, Paris, France
- Germany (2):
  - Parexel International GmbH, Berlin
  - University of Hamburg (Universitatklinikum Hamburg-Eppendorf), Hamburg
- Richmond Pharmacology (RPL), London, London Bridge, United Kingdom

IPD SHARING:
Plan to Share IPD: No